CLINICAL TRIAL: NCT06538805
Title: Dentists' Knowledge, Attitude and Practice Regarding Minimally Invasive Dentistry in Cairo and Beni-Seuf: a Cross Sectional Comparative Study
Brief Title: Dentists' Knowledge, Attitude and Practice Regarding Minimally Invasive Dentistry a Cross Sectional Comparative Study Between Two Governorates in Egypt
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Nour Alden Taha, Teaching assistant at faculty of dentistry Beni -suef university, Cairo University
Other Study IDs: MID Knowledge
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Attitude Towards Minimal Invasive Dentistry
Keywords: MID

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Minimal invasive management of dental caries — Minimal invasive management of dental caries among dentists

SUMMARY:
Some of the published researches indicate that many practicing dentists have not used the MID concepts yet in their clinics. They still use the surgical model of treatment despite the paradigm shift to the medical model. Spreading the knowledge and education about MID concepts will help in preserving more teeth structures which will be reflected on the efforts to promote the oral health in the Egyptian community. Thus the purpose of thiscross sectional study is to evaluate dentists' knowledge, attitudes, and practices regarding MID in both Cairo and Benisuef governorates.

The aim of this study is to gauge, assess and compare the knowledge, attitudes, and impact on clinical practices of dentists in Cairo and Beni-Suef governorates in Egypt regarding minimally invasive dentistry concepts.

DETAILED DESCRIPTION:
Dental caries is the most common infectious disease worldwide; approximately 36% of the world's population has carious lesions in their permanent teeth . In Egypt, dental caries is prevalent among Egyptian adolescents .In addition, dental caries, is a bacterial infectious disease that can damage teeth and restorations if microflora is not managed.

The traditional restorative method is based on G.V. Black's concept of extension for prevention. This surgical intervention pushes the tooth into a viscous circle of repeated restorations, which will eventually decrease the restoration longevity. On the contrary, minimal intervention dentistry (MID) focuses on preserving existing tooth structure and advocates a biological approach to treating dental caries. It is widely used in the dentistry curriculum to control dental cavities . The minimally invasive caries management paradigm focuses on recognizing and eliminating causal causes as well as healing carious lesions. In addition to the wide use of adhesive restorations. The MID concept utilizes new technology to create a simplified conceptual model of disease processes .

Nowadays, as a result of advancements in the field of dental restorative materials and an increased awareness of how diseases begin and progress, have paved the path for the development of minimally invasive and preventive dental caries treatment and prevention techniques . Thus,this research aims to evaluate the extent to which MID concepts for treating dental caries are popular among practicing dentists in Cairo and Benisuef.

Dental caries is a preventable infectious disease and is considered the primary cause of restorative placement and replacement . As evidence-based dentistry has developed through the years, technology has improved, and dental caries rates have reduced among the population. An innovative approach for managing dental caries emerged in the early 1970s, drawing inspiration from the principles of the medical model. This new way of thinking gave priority to conservative cavity preparations, early caries detection, adhesive restorative materials, chemotherapeutic agents, remineralization of tooth structure (fluoride), caries risk assessment, conservative cavity preparations, and tooth preservation techniques in order to minimize invasive interventions and preserve tooth structure. In the dental profession, decision-making is a challenging procedure. Numerous studies have demonstrated that a wide range of factors, including the affordability of therapy for patients, their preferences, and the training of physicians, influence this decision.

Dr. G.V. Black was the first dentist to demonstrate the treatment of dental caries using engineering principles to improve cavity preparations according to materials available at that time. The traditional restorative method is based on extension for prevention. This surgical intervention pushes the tooth into an endless circle of repeated restorations, which will eventually decrease the restoration's longevity . This traditional surgical approach prioritizes restoration material retention over sound tooth structure preservation due to the belief that caries is irreversible, patients with carious lesions are at high risk for disease progression, and restorations are often planned at the first appointment. Decisions are based on radiographic evidence, or DEJ. So Black's principles are considered an aggressive approach by modern dental standards.

The Minimally Invasive Dentistry (MID) approach focuses on early diagnosis of caries, reducing cariogenic bacteria, and minimizing invasive cavity preparations . Silver fluoridediammine was used in dentistry to establish the minimal intervention philosophy in the early 1970s . This was followed by conservative restoration, preventive resin restoration (PRR) in the 1980s, and atraumatic restorative treatment (ART) in the 1990s

. The main objectives of this medical model of caries treatment are to identify and eliminate the factors that cause caries and to repair any damage that caries causes. by synthesizing knowledge of the disease process into a simple conceptual model using new technologies .

Overall, early caries detection and activity assessment, use of diagnostic aids to classify caries depth and progression, evaluation of individual caries risk, reduction of cariogenic bacteria to lower the risk of additional demineralization, arresting of active lesions, remineralization and monitoring of non-cavitated lesions, placement of restorations using minimal cavity designs rather than replacement of defective restorations, and monitoring disease management outcomes at predetermined intervals are all included in MID .

Early diagnosis means detection of the carious lesion at early stages to be able to apply remineralization methods. Good lighting, a dry, clean field, and magnification are optimal conditions for a dentist for valid and reliable detection. The use of sharp explorers to detect initial caries is neither valid nor reliable and should be avoided .Some diagnostic tools can improve the validity and reliability of diagnoses: radiography; electrical resistance (ECM: Electrical Caries Monitor); quantitative laser and light fluorescence (QLF: Quantitative Light-induced Fluorescence); infrared laser fluorescence (IRLF); visual inspection with or without translumination; and light transmission (FOTI: Fiber Optic Trans Illumination) .

The concept of remineralization of early lesions and reduction of cariogenic bacteria can help to arrest and even reverse the mineral loss associated with caries at an early stage before cavitation takes place. Agents such as chlorhexidine, topical fluorides, hydroxy appetite and (CPP-ACP) can be applied to help in remineralization.

Minimal Cavity Preparation Design aims to remove only infected or broken areas, moving away from the surgical approach. Minimally invasive occlusal cavity preparation involves small, minimally involved dentin preparations. Some shallow lesions require minimal preparation and sealant placement. Proximal cavity designs as simple box preparations are conservative .

The Minimally Invasive Dentistry (MID) philosophy includes techniques such as the Atraumatic Restorative Technique (ART), based on removing the infected layer and maintaining the affected layer (demineralized dentin) to arrest the caries progression (Massler's theory) while using the healing potential of glass ionomer cement (GIC) to remineralize the affected dentin(Mjör and Gordan, 1999). MID also includes the lamination "sandwich" technique, which takes advantage of the combination of strong adhesion of GICs to tooth structure and the superior physical properties of the resin-based composites. The combination of the two materials, where resin composite is laminated over glass-ionomer, may offer a useful alternative in situations where the occlusal load is heavy and there is a lack of enamel to provide adhesion to resin composite . The main goals of MID are to preserve as much tooth tissue as possible and provide patients who are afraid of dental procedures with more patient-friendly care. Thus, MID can be useful in both public and private practice.

It would therefore make sense for dentists to start altering their treatment philosophies in light of growing evidence-based dentistry, new technologies, declining dental caries rates, more appropriate diagnostic procedures, increased reimbursement, and a deeper comprehension of the MID approach .Though there is evidence in the literature that dentists are utilizing MID, there has not been enough research published to determine whether or not MID use is rising.

ELIGIBILITY:
Dentists (at various levels of education, specialties and years of practice) practicing in Cairo and Beni-seuf who will choose to participate in the study.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Practicing dentist with different levels of experience in Cairo and Beni-Suef
Sampling Method: Non-Probability Sample
Enrollment: 808 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Awareness of the minimal invasive dentistry among practicing dentists in Cairo and Beni-suef | Data will be collected online over a 3-month duration
  Validated Questionnaire used in the study by (Oliveira, 2011)

SECONDARY OUTCOMES:
Comparison of knowledge, attitudes and practices between dentists from Cairo and Beni-suef regarding minimally invasive dentistry | Data will be collected online over a 3-month duration
  Validated Questionnaire used in the study by (Oliveira, 2011)